CLINICAL TRIAL: NCT00357825
Title: An 8-Week, Randomized, Double-Blind, Placebo-Controlled, Multi-Centre Study of [S,S]-Reboxetine Administered Once Daily in Patients With Fibromyalgia
Brief Title: A Trial Assessing The Effectiveness and Safety of [S,S]-Reboxetine in Patients With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6061034
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O-methyl reboxetine

INTERVENTIONS:
Drug: [S,S]-Reboxetine

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of [S,S]-Reboxetine in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* At screening patients must meet the ACR criteria for fibromyalgia (i.e. widespread pain for at least 3 months, and pain in at least 11 of 18 specific tender point sites).
* At screening and randomization, patients must have a score of >/=40mm on the Visual Analog Scale (VAS) of the Short-Form-McGill Pain Questionnaire (SF-MPQ).

Exclusion Criteria:

* Patients with other severe pain (e.g. DPN and PHN) that may confound assessment or self-evaluation of the pain associated with fibromyalgia.
* Patients with severe hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Weekly Average Pain Score from the Daily Pain Diary.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) Total Score
Patient Global Impression of Change
Short-Form 36 Health Survey (SF 36)
Sheehan Disability Scale
Medical Outcomes Study - Sleep Scale (MOS-Sleep Scale)
Quality of Sleep Score from the Daily Sleep Diary
Multidimensional Assessment of Fatigue (MAF)
Hospital Anxiety and Depression Scales (HADS)
Short-Form McGill Pain Questionnaire (SF-MPQ)
Fibromyalgia Health Assessment Questionnaire (F-HAQ)
Safety and Tolerability
Exposure Response Relationship Between Daily Dose and Daily Pain Score

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (54):
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Auburn, California
  - Pfizer Investigational Site, Orangevale, California
  - Pfizer Investigational Site, Pismo Beach, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Moline, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, Mansfield, Massachusetts
  - Pfizer Investigational Site, Wellesley Hills, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Camp Hill, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Georgetown, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Everett, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Arnold LM, Chatamra K, Hirsch I, Stoker M. Safety and efficacy of esreboxetine in patients with fibromyalgia: An 8-week, multicenter, randomized, double-blind, placebo-controlled study. Clin Ther. 2010 Aug;32(9):1618-32. doi: 10.1016/j.clinthera.2010.08.003. PMID 20974319
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061034&StudyName=A%20Trial%20Assessing%20The%20Effectiveness%20and%20Safety%20of%20%5BS%2CS%5D-Reboxetine%20in%20Patients%20With%20Fibromyalgia%0D